CLINICAL TRIAL: NCT04440540
Title: Effectiveness of Lifestyle Modification Program in Reversal of Non-alcoholic Fatty Liver Disease (NAFLD) and Reduction of Cardiovascular Risks in Moderate Obesity: A Ultrasound Attenuation Imaging-Based Study
Brief Title: Alternation of Non-alcoholic Fatty Liver Disease (NAFLD) and Cardiovascular Risks After Liftestyle Modification: A Ultrasound Attenuation Imaging-Based Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the patient recruitment was severely affected by COVID-19 pandemic
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Winnie W.C. Chu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2020.256
Record Dates: First submitted 2020-06-11; First posted 2020-06-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Ultrasound Attenuation Imaging; NAFLD; cardiovascular risk; lifestyle modification
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lifestyle modification program group (Experimental)
  Interventions: Behavioral: Dietitian led life style modification intervention
- usual care group (control) (Experimental)
  Interventions: Behavioral: Conventional care (control)

INTERVENTIONS:
Behavioral: Dietitian led life style modification intervention — lifestyle changes supervised by dietitians
  Arms: lifestyle modification program group
Behavioral: Conventional care (control) — receive routine care
  Arms: usual care group (control)

SUMMARY:
The prevalence of obesity has significantly increased over the last few decades. The excessive fat accumulation in undesired areas in obese patients may lead to various complications, such as cardiovascular diseases and Non-alcoholic fatty liver disease (NAFLD) defined by intrahepatic triglycerides (IHTG) content higher than 5.5%. In Hong Kong, the incidence rate of NAFLD is as high as approximately 13.5%, while 60.5% of obese subjects suffer from NAFLD. NAFLD is found to be a well-established risk factor for chronic kidney disease, type 2 diabetes, and cardiovascular disease. Moreover, obesity is a strong independent risk factor for development of atherosclerosis. It also plays important role in pathogenesis of dyslipidaemia, insulin resistance, hypertension. Both NAFLD and cardiovascular risks can be reversed. Lifestyle modification program(LMP) including diet control and routine exercise has been widely recommended to patients with mild to moderate obesity. It is vital to have a non-invasive, non-ionizing, low cost, accessible or widely available and yet accurate assessment tool to diagnose NAFLD and some cardiovascular risk parameters and serially monitor changes to assess the efficacy of LMP. Ultrasound meets these requirements. To the best of our knowledge there has been no prior study similar to this one. In this study, we aim to assess and validate the diagnostic accuracy of a novel ultrasound attenuation imaging method for NAFLD, and to evaluate the effectiveness of LMP in reversal of NAFLD and reduction of cardiovascular risks in moderate obesity.

A total of forty moderate obese patients with NAFLD will be recruited in this study, divided into lifestyle modification program group(n=20) and usual care group(n=20). All subjects will undergo dietary assessment based on 3-day diet record and power of food scale. Demographic data will be recorded, consisted of age, weight, height, waist circumference, BMI, and so on. Ultrasound attenuation imaging (ATI) will be performed to measure tissue attenuation coefficient so as to evaluate liver steatosis and liver fibrosis stage. Meanwhile, magnetic resonance imaging (MRI) will be carried out, which include cardiovascular risks measurement, liver proton density fat fraction (PDFF), volume quantification of abdominal white adipose tissue, liver inflammation and fibrosis assessment. Biochemistry tests will be conducted as supplementary for assessment of NAFLD and cardiovascular risks, comprising liver function test, lipid, fasting glucose, etc.

ELIGIBILITY:
Inclusion Criteria:

* With age range of 18-65 years.
* With diagnosis of NAFLD.
* BMI =27.5- 32.4kg/m2 for moderate obesity (Asian population)
* Written consent form obtained.

Exclusion Criteria:

* Other kind of hepatic diseases or under medications known to affect liver fat accumulation.
* Excessive alcohol consumption (>20g/d for men and >10g/d for women).
* Subjects using thyroid hormones, oestrogens, amiodarone, steroids, tamoxifen and beta blockers (e.g. propranolol).
* Body weight >250kgs and or/ waist circumference > 150cm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
intrahepatic triglycerides (IHTG) content | 1 year
  change of IHTG content in NAFLD assessed by ultrasound
cardiovascular risks | 1 year
  cardiovascular risks reflected by Intima-media thicknesses of both carotid arteries

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carbone S, Canada JM, Billingsley HE, Siddiqui MS, Elagizi A, Lavie CJ. Obesity paradox in cardiovascular disease: where do we stand? Vasc Health Risk Manag. 2019 May 1;15:89-100. doi: 10.2147/VHRM.S168946. eCollection 2019. PMID 31118651
- [Background] Szczepaniak LS, Nurenberg P, Leonard D, Browning JD, Reingold JS, Grundy S, Hobbs HH, Dobbins RL. Magnetic resonance spectroscopy to measure hepatic triglyceride content: prevalence of hepatic steatosis in the general population. Am J Physiol Endocrinol Metab. 2005 Feb;288(2):E462-8. doi: 10.1152/ajpendo.00064.2004. Epub 2004 Aug 31. PMID 15339742
- [Background] Wong VW, Wong GL, Yeung DK, Lau TK, Chan CK, Chim AM, Abrigo JM, Chan RS, Woo J, Tse YK, Chu WC, Chan HL. Incidence of non-alcoholic fatty liver disease in Hong Kong: a population study with paired proton-magnetic resonance spectroscopy. J Hepatol. 2015 Jan;62(1):182-9. doi: 10.1016/j.jhep.2014.08.041. Epub 2014 Sep 6. PMID 25195550
- [Background] Wong VW, Chu WC, Wong GL, Chan RS, Chim AM, Ong A, Yeung DK, Yiu KK, Chu SH, Woo J, Chan FK, Chan HL. Prevalence of non-alcoholic fatty liver disease and advanced fibrosis in Hong Kong Chinese: a population study using proton-magnetic resonance spectroscopy and transient elastography. Gut. 2012 Mar;61(3):409-15. doi: 10.1136/gutjnl-2011-300342. Epub 2011 Aug 16. PMID 21846782
- [Background] Wei JL, Leung JC, Loong TC, Wong GL, Yeung DK, Chan RS, Chan HL, Chim AM, Woo J, Chu WC, Wong VW. Prevalence and Severity of Nonalcoholic Fatty Liver Disease in Non-Obese Patients: A Population Study Using Proton-Magnetic Resonance Spectroscopy. Am J Gastroenterol. 2015 Sep;110(9):1306-14; quiz 1315. doi: 10.1038/ajg.2015.235. Epub 2015 Jul 28. PMID 26215532
- [Background] Mantovani A, Zaza G, Byrne CD, Lonardo A, Zoppini G, Bonora E, Targher G. Nonalcoholic fatty liver disease increases risk of incident chronic kidney disease: A systematic review and meta-analysis. Metabolism. 2018 Feb;79:64-76. doi: 10.1016/j.metabol.2017.11.003. Epub 2017 Nov 11. PMID 29137912
- [Background] Mantovani A, Byrne CD, Bonora E, Targher G. Nonalcoholic Fatty Liver Disease and Risk of Incident Type 2 Diabetes: A Meta-analysis. Diabetes Care. 2018 Feb;41(2):372-382. doi: 10.2337/dc17-1902. PMID 29358469
- [Background] Targher G, Byrne CD, Lonardo A, Zoppini G, Barbui C. Non-alcoholic fatty liver disease and risk of incident cardiovascular disease: A meta-analysis. J Hepatol. 2016 Sep;65(3):589-600. doi: 10.1016/j.jhep.2016.05.013. Epub 2016 May 17. PMID 27212244
- [Background] Liu Y, Zhong GC, Tan HY, Hao FB, Hu JJ. Nonalcoholic fatty liver disease and mortality from all causes, cardiovascular disease, and cancer: a meta-analysis. Sci Rep. 2019 Jul 31;9(1):11124. doi: 10.1038/s41598-019-47687-3. PMID 31366982
- [Background] Akil L, Ahmad HA. Relationships between obesity and cardiovascular diseases in four southern states and Colorado. J Health Care Poor Underserved. 2011;22(4 Suppl):61-72. doi: 10.1353/hpu.2011.0166. PMID 22102306
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Unamuno X, Gomez-Ambrosi J, Rodriguez A, Becerril S, Fruhbeck G, Catalan V. Adipokine dysregulation and adipose tissue inflammation in human obesity. Eur J Clin Invest. 2018 Sep;48(9):e12997. doi: 10.1111/eci.12997. Epub 2018 Aug 3. PMID 29995306